CLINICAL TRIAL: NCT02245308
Title: Abstinence Reinforcement Therapy (ART) for Homeless Veteran Smokers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1301-R; 1828 (Other: VA IRB)
Record Dates: First submitted 2014-09-11; First posted 2014-09-19 (Estimated); Results first posted 2019-03-07 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Tobacco Use Disorder; Homelessness
Keywords: Tobacco use cessation; Homelessness; Veterans
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation | interventions — Tobacco Use Cessation Devices; Nicotine; Nicotine Chewing Gum; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ART (Experimental): Participants assigned to this treatment arm will receive a tele-health intervention that combines guideline-based cognitive-behavioral counseling for smoking cessation, a tele-medicine clinic for access to smoking cessation aids, and an intensive behavioral therapy for smoking cessation called mobile contingency management.
  Interventions: Drug: Nicotine Patches; Behavioral: mobile contingency management (mCM); Behavioral: Smoking cessation counseling; Drug: Nicotine rescue method; Drug: Bupropion
- Control Group (Active Comparator): Participants assigned to this active control arm will be referred to VA Specialty Smoking Cessation Clinic for standard-of-care treatment, which may include group counseling, individual counseling, self-help materials, and smoking cessation aids.
  Interventions: Drug: Nicotine Patches; Behavioral: Smoking cessation counseling; Drug: Nicotine rescue method; Drug: Bupropion

INTERVENTIONS:
Drug: Nicotine Patches — Nicotine replacement therapy in the form of nicotine patches will be provided to ART group participants beginning on their smoking quit date. Nicotine patches may be provided to control group participants as part of usual care.
  Other Names: Nicoderm
Behavioral: mobile contingency management (mCM) — Mobile contingency management (mCM) is a behavioral intervention designed to provide positive reinforcement for remaining abstinent from smoking. In this intervention, participants are loaned a smart phone equipped with a videocamera and a carbon monoxide (CO) monitor. Participants are trained to upload videos of themselves taking CO readings. Any time a participant uploads a video recording that suggests abstinence (i.e., low CO reading), he/she will be provided a monetary reward.
  Arms: ART
Behavioral: Smoking cessation counseling — Smoking cessation counseling is a cognitive-behavioral treatment designed to prepare participants for a quit attempt, and to address relapse when necessary.
Drug: Nicotine rescue method — Nicotine replacement therapy in the form of nicotine gum or lozenges will be provided to ART group participants beginning on their smoking quit date. Nicotine gum or lozenges may be provided to control group participants as part of usual care.
  Other Names: Nicorette
Drug: Bupropion — Bupropion SR may be prescribed to medically eligible ART group participants beginning one week prior to quit date. Bupropion may also be prescribed to control group participants as part of usual care.
  Other Names: Zyban, Wellbutrin

SUMMARY:
The goal of this research study is to examine the effects of a treatment for helping homeless veterans who smoke to stop smoking. Participants in the study will be assigned to one of two study groups. Participants in the first group will be referred to the local Department of Veterans Affairs Medical Center's Smoking Cessation Clinic for treatment. Second group participants will receive a behavioral treatment designed to reward smokers for quitting and staying quit. These participants will also receive telephone counseling and medications for smoking cessation.

DETAILED DESCRIPTION:
Cigarette smoking is the most lethal substance use disorder in the United States in terms of morbidity and mortality. Veterans who are homeless, along with those who have mental health or substance abuse problems, are at the highest risk for nicotine dependence. Prevalence estimates for smoking among homeless Veterans are 80%. Thus, homeless Veterans are at tremendous risk for smoking related morbidity and mortality. This information suggests that smoking needs to be targeted specifically among this high risk population of smokers.

The addition of contingency management (CM) to existing evidence-based tele-health smoking cessation interventions is expected to be a cost-effective way to increase the reach of intensive smoking cessation treatment. CM is a behavioral therapy that provides positive reinforcers to individuals misusing substances contingent upon objective evidence of abstinence from substance use. Because CM requires verification of abstinence multiple times daily with a clinic-based carbon monoxide (CO) monitor, it has largely been relegated to inpatient and day treatment programs. The application of emerging smart phone technology, however, can overcome this barrier, and may be particularly well suited to homeless Veterans. The innovative smart phone application has made the use of CM for outpatient smoking cessation portable and feasible. The goal of this comparative effectiveness trial is to evaluate the effectiveness of a combined tele-health and mobile CM intervention that the investigators are calling Abstinence Reinforcement Therapy (ART). The investigators propose to screen 165 and randomize 126 homeless Veteran smokers to either:

ABSTINENCE REINFORCEMENT THERAPY (ART), a tele-health intervention that combines guideline-based cognitive-behavioral telephone (CBT) counseling, a tele-medicine clinic for access to smoking cessation aids including choice of pharmacotherapy, and intensive behavioral therapy through mCM.

VA SPECIALTY SMOKING CESSATION TREATMENT control, which includes all the elements associated with enrollment in a VA specialty smoking cessation clinic including group counseling, individual telephone counseling, self-help materials, and smoking cessation aids including choice of pharmacotherapy.

Specific aims are to:

AIM 1: Evaluate the impact of ART on rates of abstinence from cigarettes as measured by bio-verified, self-reported prolonged abstinence at post-treatment, and 3-month and 6-month post-randomization follow-ups.

AIM 2: Evaluate the relative cost-effectiveness of the ART intervention in quality adjusted life years (QALY).

AIM 3: Evaluate potential treatment mediators including self-efficacy-related mechanisms.

Supplementary AIM: To evaluate the impact of psychiatric (i.e., PTSD, depression and alcohol abuse) symptoms on treatment outcome across the two conditions.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Homeless
* Enrolled in Durham VA Medical Center for medical care
* Current smoker (at least 10 cigarettes per day)
* Willing to quit smoking in the next 30 days

Exclusion Criteria:

* Active substance dependence other than nicotine
* Uncontrolled psychotic symptoms
* Severely impaired hearing or speech (must be able to respond to telephone calls)
* Lack of interest in receiving telephone care
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean C Beckham, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five participants who signed consent were ineligible to participate in the study because they didn't meet basic eligibility criteria. One participant who signed consent was not randomized to treatment because he was unwilling to stop marijuana use prior to participating.
Groups:
- Abstinence Reinforcement Therapy: Participants assigned to this treatment arm will receive a tele-health intervention that combines:
  1. Nicotine replacement therapy in the form of nicotine patches and nicotine replacement therapy in the form of nicotine gum or lozenges provided beginning on the smoking quit date.
  2. Mobile contingency management (mCM), a behavioral intervention designed to provide positive reinforcement for remaining abstinent from smoking. In this intervention, participants are loaned a smart phone equipped with a videocamera and a carbon monoxide (CO) monitor. Participants are trained to upload videos of themselves taking CO readings, and are reinforced for readings suggesting abstinence.
  3. Smoking cessation counseling, a cognitive-behavioral treatment designed to prepare participants for a quit attempt, and to address relapse when necessary.
  4. Bupropion SR, may be prescribed to medically eligible ART group participants beginning one week prior to quit date.
Period: Overall Study
Arm/Group | Abstinence Reinforcement Therapy | Control Group
Started | 63 | 64
Completed | 63 (Using intent-to-treat analyses, i.e., missing=smoking) | 64 (Using intent-to-treat analyses, i.e., missing=smoking)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abstinence Reinforcement Therapy | Control Group | Total
Number analyzed (Participants) | 63 | 64 | 127
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.76 (10.26) | 55.72 (7.49) | 54.75 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 57 | 61 | 118
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 60 | 62 | 122
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 44 | 83
  White | 17 | 11 | 28
  More than one race | 7 | 7 | 14
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 64 | 127
Bioverified abstinent from smoking [Count of Participants; unit: Participants] | 63 | 64 | 127

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Self-reported and Bioverified Abstinent From Smoking
Description: Smoking abstinence at six months will be measured by self-report and bio-verified by salivary cotinine (a by-product of nicotine found in saliva).
Time Frame: 6 months
Population: All participants who were randomized to treatment were included in the final analysis of bioverified abstinence, using an intent-to-treat sample where missing = smoking
Measure: Count of Participants; unit: Participants
Arm/Group | Abstinence Reinforcement Therapy | Control Group
Number analyzed (Participants) | 63 | 64
Participants | 13 | 5

2. Secondary Outcome: Intervention Delivery Costs
Description: Intervention delivery costs (including medication costs, supplies, and incentive pay for abstinence) will be evaluated for treatment and control group.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: dollars
Arm/Group | Abstinence Reinforcement Therapy | Control Group
Number analyzed (Participants) | 63 | 64
dollars | 618.35 (180.02) | 226.00 (0)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over a one year period.
Description: clinicaltrials.gov definitions were used.
Arm/Group | Abstinence Reinforcement Therapy | Control Group
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/63 | 1/64
Other Adverse Events (participants affected / at risk) | 15/63 | 18/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abstinence Reinforcement Therapy (N=63) | Control Group (N=64)
High blood pressure (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abstinence Reinforcement Therapy (N=63) | Control Group (N=64)
Nausea or upset stomach (Gastrointestinal disorders) | 3 (3) | 3 (3)
Skin irritation or rash (Skin and subcutaneous tissue disorders) | 6 (8) | 10 (15) — Due to nicotine patch use
Sleep difficulties or nightmares (General disorders) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT02245308/Prot_SAP_000.pdf